CLINICAL TRIAL: NCT07403045
Title: Effects of McGill Strengthening Exercises Program With and Without Integrated Neuromuscular Inhibition Technique on Pain, Range of Motion and Function in Patients With Piriformis Syndrome
Brief Title: McGill Strengthening With and Without Integrated Neuromuscular Inhibition Technique in Piriformis Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0176
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Piriformis Syndrome
Keywords: integrated neuromuscular inhibition technique; McGill exercises; pain; physical functional performance; piriformis syndrome; range of motion; trigger points
MeSH Terms: conditions — Piriformis Muscle Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- McGill strengthening exercises program with integrated neuromuscular inhibition technique (Experimental)
  Interventions: Other: McGill strengthening exercises program; Other: Integrated neuromuscular inhibition technique; Other: Standardized physiotherapy treatment
- McGill strengthening exercises program (Active Comparator)
  Interventions: Other: McGill strengthening exercises program; Other: Standardized physiotherapy treatment

INTERVENTIONS:
Other: McGill strengthening exercises program — These exercises were divided into 3 phases, each lasting 2 weeks. Patients performed 4 repetitions of each exercise during 1st and 2nd week at each hospital visit. Then, increased by 4 repetitions every 2 weeks for up to 6 weeks. These exercises were performed with a maximum of 12 repetitions with a 1-minute of rest interval between each exercise. These exercises were performed by patients at each clinical visit, 3 days per week for total of 6 weeks.
Other: Integrated neuromuscular inhibition technique — This technique was applied at piriformis muscle. The procedure was repeated 3 times for up to 10 minutes at each clinical visit. This intervention was performed 3 days per week for total of 6 weeks.
  Arms: McGill strengthening exercises program with integrated neuromuscular inhibition technique
Other: Standardized physiotherapy treatment — These exercises were performed by patients at the end of each hospital visit (3 days per week for total of 6 weeks) and also at home twice a week during the 2 months follow-up period after treatment ends.
  1. Continuous-mode ultrasound therapy was applied at a frequency of 1 MHz and an intensity of 1.0 W/cm² for 3 minutes to the tender or trigger points on the posterior aspect of the pelvis.
  2. A hydrocollator pack (40°C) was applied for 10 minutes at lumbopelvic region.
  3. Piriformis, hamstring/calf stretching was performed progressively in phases.
     * Phase 1 consists of weeks 1 and 2 with 1 set of 3 repetitions with 30 seconds hold per day.
     * Phase 2 consists of weeks 3 and 4 with 2 sets of 3 repetitions with 30 seconds hold per day.
     * Phase 3 consists of weeks 5 and 6 with 2 sets of 3 repetitions with 30 seconds hold twice per day.
     * Follow-up period consists of 2 sets of 3 repetitions with 30 seconds hold twice per day.

SUMMARY:
The study was conducted to determine the effects of McGill strengthening exercises program with and without integrated neuromuscular inhibition technique on pain, range of motion and function in patients with piriformis syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Both genders with age ranged from 25 and 45 years
* Sedentary
* Non-traumatic
* Idiopathic
* External tenderness near the greater sciatic notch
* Pain for more than 1 month's duration
* NPRS ranging from >3 to ≤ 6
* Positive results on three of the following five tests:

  1. FAIR
  2. Beatty
  3. Laségue
  4. Pace
  5. Freiberg

Exclusion Criteria:

* Acute low back pain and/or acute lumbar radiculopathy
* History of Stroke or any other neurological disorders
* Recent buttock trauma
* Inflammatory, infectious or tumor diseases
* Severe vascular disease
* Osteoporosis
* Pregnancy

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | From enrollment to 6 weeks of intervention with follow-up at 14 weeks.
  Numeric Pain Rating Scale (NPRS) was used to assess the patient's pain intensity. This scale ranges from 0 to 10, where 0 indicates "no pain" and 10 indicates "worst pain.

SECONDARY OUTCOMES:
Range of Motion (Hip Abduction) | From enrollment to 6 weeks of intervention with follow-up at 14 weeks.
  The universal goniometer was used to assess hip abduction range of motion.
Range of Motion (Hip Internal Rotation) | From enrollment to 6 weeks of intervention with follow-up at 14 weeks.
  The universal goniometer was used to assess hip internal rotation range of motion.
Lower Extremity Functional Scale | From enrollment to 6 weeks of intervention with follow-up at 14 weeks.
  Lower Extremity Functional Scale was used to assess the patient's functional status. Maximum score of this scale is 80. The greater the score, the lower the disability.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, PhD, Study Director — Riphah International University
Locations (1):
- Mumtaz Bakhtawar Memorial Trust Hospital, Mustafa Town, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nazlikul H, Ural FG, Ozturk GT, Ozturk ADT. Evaluation of neural therapy effect in patients with piriformis syndrome. J Back Musculoskelet Rehabil. 2018;31(6):1105-1110. doi: 10.3233/BMR-170980. PMID 30010101
- [Background] Jamaly A, Mohsenifar H, Amiri A. The effects of dry needling in combination with physical therapy on improvement of pain and hip internal rotation range in patients with piriformis syndrome. Journal of Clinical Physiotherapy Research. 2018;3(3):118-22.
- [Background] Awan WA, Babur MN, Ali S, Janjua U. The effectiveness of electrotherapy with manual therapy in the treatment of piriformis syndrome. Int J Rehabil Sci. 2018;1(1):16-9.
- [Background] Laha K, Sarkar B, Kumar P, Patel L, Sarkar N. Efficacy of hip abductor and extensor strengthening on pain, strength and lower extremity function in piriformis syndrome: a randomized clinical trial. Int J Health Sci Res. 2018;8(9):80-.
- [Background] Velappanchavadi C. Effectiveness of muscle energy technique versus stretching in subjects with piriformis syndrome. Int J Physiother Res. 2019;7(5):3252-56.
- [Background] Alarab A, Unver F. Stretching exercise versus tissue mobilization technique in piriformis syndrome. European Journal of Medical and Health Sciences. 2020;2(6).
- [Background] Kutty NN, Siddeeque S, Tamphaibema H, Othayoth N, Bineesh CP. Effect of Muscle Energy Technique with Deep Friction Massage on Pain, Disability and Internal Rotation Range of Motion of Hip Joint in Individuals with Piriformis Syndrome. Indian Journal of Physiotherapy & Occupational Therapy. 2020 Jan 1;14(1).
- [Background] Athawale VK, Jethwani D, Qureshi MD, Dadgal R. Combined Effect of Neural Tissue Mobilization and Deep Friction Massage in Piriformis Syndrome: A Research Protocol. Indian Journal of Forensic Medicine & Toxicology. 2021 Apr 1;15(2).
- [Background] Chaudhary S, Sheikh M, Chaudhary NI, Ambad R, Bankar N. Effect of neural tissue mobilization in combination with ultrasonic therapy verses ultrasonic therapy in deep gluteal syndrome-a comparative study.
- [Background] RAZA H, ARSLAN HR, IQBAL A, HAMID MF, WASEEM A, MANZOOR S. Comparison Of Gluteal Muscle Strengthening Versus Conventional Isometrics In Pain Management Of Piriformis Syndrome. Age (years). 2021 Nov 1;50(5.79):45-31.
- [Background] Roy S, Solanki N, Phd AC. Effectiveness of muscle energy technique versus static stretching in subject with tight piriformis in male office going subjects: a randomized clinical trial. IJRAR-International J Res Anal Rev. 2022;9(3):295-321.
- [Background] Idrees KI, Khan KH, Sharif KH, Ahmad KH, Rahman HA, Fahad FA. Efficacy Of Hip Abductors Strengthening As Compared To Piriformis Muscle Stretching In Improving Lower Extremity Function In Patients With Piriformis Syndrome. Pakistan Journal of Medical & Health Sciences. 2022 Sep 16;16(07):721.
- [Background] Ahmad N, Akram MJ, Hussain H, Imtiaz I, Khan N, Qi L. Effectiveness of post facilitation stretch technique versus myofascial release in piriformis syndrome: A Randomized controlled trial. Rawal Medical Journal. 2022 Nov 12;47(4):936.
- [Background] Shahzadi B, Taj S, Nawaz S, Hamid I, Talpur MA, Hussain SA, Sajjad AG, Kiyani M. Sacroiliac joint manipulation helps to improve pain pressure threshold in chronic piriformis syndrome: a 6-week randomized controlled trial. The Rehabilitation Journal. 2023 Mar 31;7(01):476-82.
- [Background] Ergezen G, Sahin M. Comparison of self-myofascial release and stretching exercises in individuals with piriformis syndrome: a randomised controlled trial. International Journal of Therapy And Rehabilitation. 2023 Nov 2;30(11):1-0.
- [Background] Aroob Z, Bashir MS, Noor R, Ikram M, Ramzan F, Naseer A, Sabir N. Comparative effects of fascial distortion model with and without neuromuscular inhibition technique on pain, range of motion and quality of life in patients with piriformis syndrome. Disabil Rehabil. 2025 May;47(9):2378-2383. doi: 10.1080/09638288.2024.2395456. Epub 2024 Sep 3. PMID 39224057
- [Background] Ilyas N, Jamil A, Akram S, Ilyas R, Afzal Z, Akram A. Comparative effects of hold relax with agonist contraction and active release therapy on pain, functional disability and sleep quality in piriformis syndrome.
- [Background] Danazumi MS, Yakasai AM, Ibrahim AA, Shehu UT, Ibrahim SU. Effect of integrated neuromuscular inhibition technique compared with positional release technique in the management of piriformis syndrome. J Osteopath Med. 2021 May 31;121(8):693-703. doi: 10.1515/jom-2020-0327. PMID 34049428
- [Background] Rehman AU, Khan LG, Khalid M, Mumtaz U, Akhtar H, Gondal A, Waris S. Comparison of active release technique and post isometric relaxation in patients with piriformis syndrome. Pakistan Journal of Medical & Health Sciences. 2022 Jun 18;16(05):683-.
- [Background] Kanwal R, Khan J, Awan WA, Khan R, Malik S. STRETCHING EXERCISES VERSUS DEEP FRICTION MASSAGE FOR THE MANAGEMENT OF PIRIFORMIS SYNDROME: soi: 21-2017/re-trjvol02iss02p65. The Rehabilitation Journal. 2018 Dec 31;2(02):65-9.
- [Background] Hernándeza DM, Pérez SM, Ardón FB, Núñez CL, Moreno JG. Effectiveness of neurodynamic mobilization and MCGILL-type strengthening exercises in patients with piriformis syndrome: study protocol for a randomized controlled trial. Physical Rehabilitation and Recreational Health Technologies. 2024 Jun 1;9(3):188-200.
- [Background] Nambi G, Dusad G. Effect of reciprocal inhibition and post isometric relaxation; types of muscle energy technique in piriformis syndrome.-a comparative study. Phys Med Rehabil Res. 2018 Apr 2;3(1):1-5.
- [Background] Shahzad M, Rafique N, Shakil-Ur-Rehman S, Ali Hussain S. Effects of ELDOA and post-facilitation stretching technique on pain and functional performance in patients with piriformis syndrome: A randomized controlled trial. J Back Musculoskelet Rehabil. 2020;33(6):983-988. doi: 10.3233/BMR-181290. PMID 32894238